CLINICAL TRIAL: NCT01379703
Title: Multicountry, Multicenter Post-Marketing Observational Study of Clinical, Biological and Virological Outcomes, Compliance and Tolerability of Kaletra® in Routine Clinical Use
Acronym: KaleEAST
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: PMOS-EAST-04-1
Record Dates: First submitted 2011-06-22; First posted 2011-06-23 (Estimated); Results first posted 2011-09-12 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: HIV-1 Patients
Keywords: HIV-1 infected patients; Protease inhibitor; Kaletra®

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single patients group: Single HIV-1 infected patients group

SUMMARY:
KaleEAST is a non-interventional, post-marketing observational study (PMOS) in which lopinavir/ritonavir is prescribed in the usual manner in accordance with the terms of the local marketing authorization with regards to dose, population and indication. No additional procedures (other than the standard of care) are to be applied to the patients.

The KaleEAST PMOS was conducted in a prospective, single-arm, multicountry, multicenter format. The study was carried out in two (2) parts: the first part was initiated in 2004 with the lopinavir/ritonavir capsule formulation, the second part started in 2006 after the lopinavir/ritonavir tablets had become available in the participating countries.

The aim of this post-marketing observational study was to obtain further data on clinical, biological, and virological outcomes, compliance and tolerability of Kaletra®-containing regimen during routine clinical use in the participating countries.

DETAILED DESCRIPTION:
As this study is observational in nature, subject follow-up was not specified by the protocol but was left to the judgment of each physician within the 18 months period, which defines the survey for each participant. For indicative purposes, follow-up of each participant should enable approximately 7 visits during this period. These visits will take place at average intervals of 3 months, apart from the first visit following inclusion (usually at the end of the first treatment month) and apart from visits required because of intercurrent events. Participant visits were assigned as follows: Baseline/Day 0 (start of lopinavir/ritonavir treatment), Month 1 (day 1 to day 45), Month 3 (day 46 to day 136), Month 6 (day 137 to day 228), Month 9 (day 229 to day 319), Month 12 (day 320 to day 410), Month 15 (day 411 to day 501), Month 18 (day 502 to day 593). Each participant is planned to be observed during his/her lopinavir/ritonavir capsule containing treatment regimen for a maximum period of 18 months, and each participant is planned to be observed during his/her lopinavir/ritonavir tablet containing treatment regimen for a maximum period of 9 months.

ELIGIBILITY:
Inclusion Criteria:

Patients infected by HIV-1 infection who are either:

* Antiretroviral treatment (ART) naive or
* Had failed or had been intolerant to one previous combined antiretroviral treatment (cART), not including a Protease inhibitor (PI) (first-line pretreated without a Protease inhibitor) or
* Had failed or had been intolerant to one previous antiretroviral treatment ART, including one Protease inhibitor (first-line pretreated with a Protease Inhibitor).

A ritonavir-boosted Protease inhibitor PI is considered as treatment with one Protease inhibitor PI.

Exclusion Criteria:

* Treatment with drugs at risk for interactions with lopinavir/ritonavir
* Uncontrolled AIDS defining disease
* Two or more previous Protease inhibitors (PIs)
* Participation in another study or clinical trial

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: KaleEAST is non-interventional, observational study in which Kaletra® is prescribed in the usual manner in accordance with the terms of the local marketing authorization with regard to dose, population and indication.
Sampling Method: Non-Probability Sample
Enrollment: 2288 (Actual)
Dates: Start 2004-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maja Hojnik, MD, PhD, Study Director — Abbott International
Locations (103):
- Czechia (7):
  - Site Ref # / Investigator 57102, Brno
  - Site Ref # / Investigator 57054, České Budějovice
  - Site Ref # / Investigator 57055, Hradec Králové
  - Site Ref # / Investigator 57056, Ostrava
  - Site Ref # / Investigator 57052, Pilsen
  - Site Ref # / Investigator 5344, Prague
  - Site Ref # / Investigator 57053, Ústí nad Labem
- Site Ref # / Investigator 7576, Tbilisi, Georgia
- Israel (6):
  - Site Ref # / Investigator 57050, Beersheba
  - Site Ref # / Investigator 57048, Haifa
  - Site Ref # / Investigator 57049, Jerusalem
  - Site Ref # / Investigator 6124, Kfar Saba
  - Site Ref # / Investigator 57047, Rehovot
  - Site Ref # / Investigator 57051, Tel Litwinsky
- Site Ref # / Investigator 7578, Riga, Latvia
- Site Ref # / Investigator 6127, Vilnius, Lithuania
- Poland (10):
  - Site Ref # / Investigator 6190, Bialystok
  - Site Ref # / Investigator 56885, Bydgoszcz
  - Site Ref # / Investigator 56887, Chorzów
  - Site Ref # / Investigator 56883, Gdansk
  - Site Ref # / Investigator 56888, Krakow
  - Site Ref # / Investigator 56889, Lodz
  - Site Ref # / Investigator 56884, Poznan
  - Site Ref # / Investigator 56886, Szczecin
  - Site Ref # / Investigator 56882, Warsaw
  - Site Ref # / Investigator 56890, Wroclaw
- Romania (8):
  - Site Ref # / Investigator 57064, Brasov
  - Site Ref # / Investigator 6194, Bucharest
  - Site Ref # / Investigator 57062, Bucharest
  - Site Ref # / Investigator 57063, Constanța
  - Site Ref # / Investigator 57067, Craiova
  - Site Ref # / Investigator 57068, Iași
  - Site Ref # / Investigator 57065, Târgu Mureş
  - Site Ref # / Investigator 57066, Timișoara
- Russia (58):
  - Site Ref # / Investigator 57022, Barnaul
  - Site Ref # / Investigator 56918, Chelyabinsk
  - Site Ref # / Investigator 56963, Chita
  - Site Ref # / Investigator 56921, Irkutsk
  - Site Ref #/Investigator 57104, Irkutsk
  - Site Ref # / Investigator 57028, Ivanovo
  - Site Ref # / Investigator 57036, Izhevsk
  - Site Ref # / Investigator 56945, Kaliningrad
  - Site Ref # / Investigator 56909, Kazan'
  - Site Ref # / Investigator 57037, Kemerovo
  - Site Ref #/Investigator 57105, Kemerovo
  - Site Ref # / Investigator 56948, Khabarovsk
  - Site Ref # / Investigator 56932, Khanty-Mansiysk
  - Site Ref #/Investigator 57107, Kirov
  - Site Ref # / Investigator 57030, Kostroma
  - Site Ref # / Investigator 56943, Krasnodar
  - Site Ref # / Investigator 56928, Krasnoyarsk
  - Site Ref #/Investigator 57106, Krasnoyarsk
  - Site Ref # / Investigator 57021, Kurgan
  - Site Ref # / Investigator 57025, Lipetsk
  - Site Ref # / Investigator 56944, Magnitogorsk
  - Site Ref # / Investigator 56904, Moscow
  - Site Ref # / Investigator 6209, Moscow
  - Site Ref # / Investigator 56902, Moscow
  - Site Ref # / Investigator 57024, Murmansk
  - Site Ref # / Investigator 56907, Nizhny Novgorod
  - Site Ref # / Investigator 56964, Noril'sk
  - Site Ref # / Investigator 56929, Novokuznetsk
  - Site Ref # / Investigator 56942, Novosibirsk
  - Site Ref # / Investigator 56926, Noyabrsk
  - Site Ref # / Investigator 56915, Orenburg
  - Site Ref # / Investigator 57031, Orenburg
  - Site Ref # / Investigator 56930, Perm
  - Site Ref # / Investigator 56911, Rostov-on-Don
  - Site Ref # / Investigator 57033, Saint Petersburg
  - Site Ref # / Investigator 56906, Saint Petersburg
  - Site Ref # / Investigator 56905, Saint Petersburg
  - Site Ref # / Investigator 56920, Saint Petersburg
  - Site Ref # / Investigator 57038, Saint Petersburg
  - Site Ref # / Investigator 56931, Samara
  - Site Ref # / Investigator 56913, Saratov
  - Site Ref # / Investigator 56908, Surgut
  - Site Ref # / Investigator 56962, Tolyatti
  - Site Ref # / Investigator 57034, Tula
  - Site Ref # / Investigator 56947, Tver'
  - Site Ref # / Investigator 57035, Tver'
  - Site Ref # / Investigator 56910, Tyumen
  - Site Ref # / Investigator 56919, Tyumen
  - Site Ref # / Investigator 57029, Ufa
  - Site Ref # / Investigator 56949, Ulan-Ude
  - Site Ref # / Investigator 56914, Ulyanovsk
  - Site Ref # / Investigator 57027, Vladimir
  - Site Ref # / Investigator 56916, Volgograd
  - Site Ref #/Investigator 57103, Vologda
  - Site Ref # / Investigator 56946, Yakutsk
  - Site Ref # / Investigator 57026, Yaroslavl
  - Site Ref # / Investigator 56923, Yekaterinburg
  - Site Ref # / Investigator 56903, Yekaterinburg
- Site Ref # / Investigator 7579, Belgrade, Serbia
- Site Ref # / Investigator 6208, Bratislava, Slovakia
- Site Ref # / Investigator 6199, Ljubljana, Slovenia
- Ukraine (8):
  - Site Ref # / Investigator 57042, Dnipro
  - Site Ref # / Investigator 57043, Donetsk
  - Site Ref # / Investigator 57045, Kyiv
  - Site Ref # / Investigator 6191, Kyiv
  - Site Ref # / Investigator 57046, Kyiv
  - Site Ref # / Investigator 57044, Mykolaiv
  - Site Ref # / Investigator 57039, Odesa
  - Site Ref # / Investigator 57040, Simferopol

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was carried out in two parts. The first part was initiated in 2004 with the lopinavir/ritonavir capsule formulation (Part I) and the second part (Part II) started in 2006 after the tablet formulation became available in participating countries.
Groups:
- Tablets and Capsules or Oral Solution: HIV-1 infected participants who received both tablet and capsule formulations or oral solution.
- Capsule Formulation: Participants who received the capsule formulation (only) of lopinavir/ritonavir during Part I or Part II of the study.
- Tablet Formulation: Participants who received the tablet formulation (only) of lopinavir/ritonavir during Parts I or II of the study.
Period: Study Start Through 9 Months
Arm/Group | Tablets and Capsules or Oral Solution | Capsule Formulation | Tablet Formulation
Started | 66 (Participants taking lopinavir/ritonavir tablets/capsules or oral solution during the study (66/2288)) | 1206 (Participants taking the lopinavir/ritonavir capsule formulation (only) during study (1206/2288)) | 1016 (Participants taking the lopinavir/ritonavir tablet formulation (only) during study (1016/2288))
Completed | 62 | 1084 (Participants taking the capsule formulation were followed for an additional 9 months (up to 18 mos).) | 873
Not Completed | 4 | 122 | 143
Not completed — Lost to Follow-up | 2 | 61 | 104
Not completed — Adverse Event | 0 | 14 | 10
Not completed — Withdrawal by Subject | 0 | 6 | 1
Not completed — Treatment Failure | 0 | 2 | 2
Not completed — Patient Noncompliance | 0 | 0 | 1
Not completed — Tuberculosis/TB treatment | 0 | 4 | 0
Not completed — Medication not available | 0 | 2 | 1
Not completed — Poor general condition | 0 | 1 | 0
Not completed — Increased triglycerides | 0 | 1 | 0
Not completed — Reason unknown | 2 | 31 | 24
Period: 9 Months Through 18 Months
Arm/Group | Tablets and Capsules or Oral Solution | Capsule Formulation | Tablet Formulation
Started | 0 (Participants in this subgroup were followed for 9 months.) | 1084 (Participants taking the capsule formulation were followed for an additional 9 months (up to 18 mos).) | 0 (Participants in this subgroup were followed for 9 months.)
Completed | 0 | 854 | 0
Not Completed | 0 | 230 | 0
Not completed — Lost to Follow-up | 0 | 178 | 0
Not completed — Withdrawal by Subject | 0 | 11 | 0
Not completed — Adverse Event | 0 | 6 | 0
Not completed — Treatment failure | 0 | 5 | 0
Not completed — Patient Noncompliance | 0 | 4 | 0
Not completed — Tuberculosis/TB treatment | 0 | 2 | 0
Not completed — Fatigue | 0 | 1 | 0
Not completed — Reason Unknown | 0 | 23 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Study Population: HIV-1 infected participants who received lopinavir/ritonavir (any formulation) during any part of the study.
Arm/Group | Total Study Population
Number analyzed (Participants) | 2288
Age Continuous [Mean (Standard Deviation); unit: years] | 32.6 (11.0)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 867
  Male | 1419
  Data not reported | 2
Region of Enrollment [Number; unit: participants]
  Serbia | 149
  Czech Republic | 107
  Slovenia | 123
  Slovakia | 26
  Poland | 381
  Ukraine | 266
  Romania | 422
  Lithuania | 3
  Russian Federation | 644
  Israel | 139
  Georgia | 10
  Latvia | 18

OUTCOME MEASURES:

1. Primary Outcome: CD4 Count
Description: CD4 lymphocyte count is a measure of a participant's immunologic health. Participants' CD4-positive (CD4+) T-lymphocyte counts were assessed by measuring the number of CD4+ cells at baseline.
Time Frame: Baseline
Population: Mean CD4 count is based on number of participants in each group who had CD4 count results at Baseline.
Measure: Mean (Standard Deviation); unit: cells per mm³
Groups:
- Total Study Population: HIV-1 infected participants who received any formulation of lopinavir/ritonavir during Parts I or II of the study (including 66 participants who received both tablet and capsule formulations, or oral solution).
Arm/Group | Total Study Population | Capsule Formulation | Tablet Formulation
Number analyzed (Participants) | 2220 | 1165 | 993
cells per mm³
  Mean CD4 count | 229.9 (194.2) | 208.8 (187.2) | 246.8 (194.8)

2. Primary Outcome: Changes in CD4 Count
Description: Increases in CD4 count are a biomarker for antiretroviral treatment effectiveness in restoring immunologic function. Changes in participants' CD4-positive (CD4+) T-lymphocyte counts were assessed by measuring the change from Baseline in the number of CD4+ cells at scheduled study visits.
Time Frame: Baseline to 1 month
Population: Change from baseline analysis is based on participants with CD4 count results available at 1 month.
Measure: Mean (Standard Deviation); unit: cells per mm³
Arm/Group | Total Study Population | Capsule Formulation | Tablet Formulation
Number analyzed (Participants) | 670 | 348 | 293
cells per mm³
  Mean CD4 count at 1 month | 288.7 (185.1) | 277.1 (195.7) | 296.1 (172.1)
  Change in CD4 count | 60.3 (137.4) | 54.9 (158.3) | 70.6 (113.8)

3. Primary Outcome: Changes in CD4 Count
Description: as for outcome 2
Time Frame: Baseline to 3 months
Population: Change from baseline analysis is based on participants with CD4 count results available at 3 months.
Measure: Mean (Standard Deviation); unit: cells per mm³
Arm/Group | Total Study Population | Capsule Formulation | Tablet Formulation
Number analyzed (Participants) | 1633 | 838 | 738
cells per mm³
  Mean CD4 count at 3 months | 323.9 (219.3) | 310.1 (227.9) | 332.4 (206.7)
  Change in CD4 count | 94.5 (162.9) | 97.7 (188.7) | 93.2 (123.9)

4. Primary Outcome: Changes in CD4 Count
Description: as for outcome 2
Time Frame: Baseline to 6 months
Population: Change from baseline analysis is based on participants with CD4 count results available at 6 months.
Measure: Mean (Standard Deviation); unit: cells per mm³
Arm/Group | Total Study Population | Capsule Formulation | Tablet Formulation
Number analyzed (Participants) | 1533 | 780 | 699
cells per mm³
  Mean CD4 count at 6 months | 361.5 (248.9) | 333.4 (219.8) | 382.0 (271.7)
  Change in CD4 count | 124.4 (197.6) | 117.1 (182.5) | 131.6 (216.0)

5. Primary Outcome: Changes in CD4 Count
Description: as for outcome 2
Time Frame: Baseline to 9 months
Population: Change from baseline analysis is based on participants with CD4 count results available at 9 months.
Measure: Mean (Standard Deviation); unit: cells per mm³
Arm/Group | Total Study Population | Capsule Formulation | Tablet Formulation
Number analyzed (Participants) | 1410 | 713 | 645
cells per mm³
  Mean CD4 count at 9 months | 384.1 (221.4) | 363.5 (222.2) | 395.0 (209.0)
  Change in CD4 count | 151.5 (174.4) | 144.8 (191.7) | 156.0 (151.5)

6. Primary Outcome: Changes in CD4 Count
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: Only participants receiving lopinavir/ritonavir capsules were planned to be followed past 9 months. Change from baseline analysis is based on participants receiving capsule formulation with CD4 count results available at 12 months.
Measure: Mean (Standard Deviation); unit: cells per mm³
Groups:
- Capsule Formulation: Participants who received the capsule formulation of lopinavir/ritonavir during Part 1 or Part II of the study.
Arm/Group | Capsule Formulation
Number analyzed (Participants) | 729
cells per mm³
  Mean CD4 count at 12 months | 392.0 (216.5)
  Change in CD4 count | 170.4 (201.7)

7. Primary Outcome: Changes in CD4 Count
Description: as for outcome 2
Time Frame: Baseline to 15 months
Population: Only participants receiving lopinavir/ritonavir capsules were planned to be followed past 9 months. Change from baseline analysis is based on participants receiving capsule formulation with CD4 count results available at 15 months.
Measure: Mean (Standard Deviation); unit: cells per mm³
Arm/Group | Capsule Formulation
Number analyzed (Participants) | 701
cells per mm³
  Mean CD4 count at 15 months | 412.6 (240.5)
  Change in CD4 count | 194.8 (228.5)

8. Primary Outcome: Changes in CD4 Count
Description: as for outcome 2
Time Frame: Baseline to 18 months
Population: Only participants receiving lopinavir/ritonavir capsules were planned to be followed past 9 months. Change from baseline analysis is based on participants receiving capsule formulation with CD4 count results available at 18 months.
Measure: Mean (Standard Deviation); unit: cells per mm³
Arm/Group | Capsule Formulation
Number analyzed (Participants) | 599
cells per mm³
  Mean CD4 count at 18 months | 429.7 (249.4)
  Change in CD4 count | 222.2 (228.7)

9. Primary Outcome: Viral Load
Description: Viral load is a direct measure of the viral burden by providing a count of the number of HIV-RNA copies in blood (plasma). The number of HIV-RNA copies in the blood was measured at baseline.
Time Frame: Baseline
Population: Mean viral load is based on number of participants in each group who had laboratory results for viral load at baseline.
Measure: Mean (Standard Deviation); unit: Log10 copies per ml
Arm/Group | Total Study Population | Capsule Formulation | Tablet Formulation
Number analyzed (Participants) | 1572 | 739 | 781
Log10 copies per ml
  Mean viral load | 4.44 (1.26) | 4.49 (1.17) | 4.43 (1.31)

10. Primary Outcome: Viral Load
Description: Viral load (number of HIV-RNA copies in the blood) was measured at baseline and scheduled study visits. A decrease in viral load is a measure used to assess the effectiveness of antiviral treatments.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: Log10 copies per ml
Arm/Group | Total Study Population | Capsule Formulation | Tablet Formulation
Number analyzed (Participants) | 420 | 218 | 175
Log10 copies per ml | 3.28 (1.08) | 3.42 (1.07) | 3.19 (1.04)

11. Primary Outcome: Viral Load
Description: as for outcome 10
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Log10 copies per ml
Arm/Group | Total Study Population | Capsule Formulation | Tablet Formulation
Number analyzed (Participants) | 995 | 469 | 478
Log10 copies per ml | 2.69 (1.00) | 2.86 (0.97) | 2.54 (1.00)

12. Primary Outcome: Viral Load
Description: as for outcome 10
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Log10 copies per ml
Arm/Group | Total Study Population | Capsule Formulation | Tablet Formulation
Number analyzed (Participants) | 1093 | 506 | 544
Log10 copies per ml | 2.40 (0.89) | 2.62 (0.88) | 2.21 (0.84)

13. Primary Outcome: Viral Load
Description: as for outcome 10
Time Frame: 9 months
Population: Change from baseline analysis is based on last observation carried forward for total study population (N=1341) and tablet formulation group (N=677).
Measure: Mean (Standard Deviation); unit: Log10 copies per ml
Arm/Group | Total Study Population | Capsule Formulation | Tablet Formulation
Number analyzed (Participants) | 918 | 406 | 471
Log10 copies per ml
  Mean viral load at 9 months | 2.41 (0.96) | 2.65 (1.02) | 2.24 (0.88)
  Change in viral load | -2.05 (1.42) | NA (NA) — Change from baseline LOCF analysis for participants receiving capsule formulation was performed at 18 months. | -2.21 (1.44)

14. Primary Outcome: Viral Load
Description: as for outcome 10
Time Frame: 12 months
Population: Only participants receiving lopinavir/ritonavir capsules were planned to be followed past 9 months.
Measure: Mean (Standard Deviation); unit: Log10 copies per ml
Arm/Group | Capsule Formulation
Number analyzed (Participants) | 444
Log10 copies per ml | 2.54 (0.92)

15. Primary Outcome: Viral Load
Description: as for outcome 10
Time Frame: 15 months
Population: Only participants receiving lopinavir/ritonavir capsules were planned to be followed past 9 months.
Measure: Mean (Standard Deviation); unit: Log10 copies per ml
Arm/Group | Capsule Formulation
Number analyzed (Participants) | 432
Log10 copies per ml | 2.49 (0.92)

16. Primary Outcome: Viral Load
Description: as for outcome 10
Time Frame: 18 months
Population: Only participants receiving lopinavir/ritonavir capsules were planned to be followed past 9 months. Change from baseline analysis is based on last observation carried forward (N=660).
Measure: Mean (Standard Deviation); unit: Log10 copies per ml
Arm/Group | Capsule Formulation
Number analyzed (Participants) | 413
Log10 copies per ml
  Mean viral load at 18 months | 2.35 (0.84)
  Change in viral load | -1.95 (1.42)

17. Primary Outcome: Laboratory Parameter Blood Glucose
Description: Blood glucose laboratory values were assessed at baseline and scheduled study visits. Normal ranges are based on the standards for individual facilities in each country.
Time Frame: Baseline, 9 months, 18 months
Population: Analysis was based on participants with laboratory values at each time point. Only participants receiving lopinavir/ritonavir capsules were planned to be followed after 9 months.
Measure: Mean (Standard Deviation); unit: millimoles per liter
Arm/Group | Total Study Population | Capsule Formulation | Tablet Formulation
Number analyzed (Participants) | 1831 | 875 | 899
millimoles per liter
  Baseline | 4.87 (2.05) | 4.89 (2.83) | 4.85 (0.86)
  9 months | 4.92 (1.42) | 4.87 (1.38) | 4.99 (1.49)
  18 months | NA (NA) — Only participants who received lopinavir/ritonavir capsules were planned to be followed past 9 months. | 5.07 (2.64) | NA (NA) — Only participants who received lopinavir/ritonavir capsules were planned to be followed past 9 months.

18. Primary Outcome: Laboratory Parameter Transaminases
Description: Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) laboratory values were assessed at baseline and scheduled study visits. Normal ranges are based on the standards for individual facilities in each country.
Time Frame: Baseline, 9 months, 18 months
Population: Analysis was based on participants with laboratory values at each time point. Only participants receiving lopinavir/ritonavir capsules were planned to be followed past 9 months.
Measure: Mean (Standard Deviation); unit: international units per liter
Arm/Group | Total Study Population | Capsule Formulation | Tablet Formulation
Number analyzed (Participants) | 2288 | 1206 | 1016
international units per liter
  AST - Baseline | 38.9 (37.1) | 36.8 (32.1) | 41.4 (42.4)
  AST - 9 months | 35.2 (33.0) | 34.8 (29.6) | 36.0 (36.9)
  AST - 18 months | NA (NA) — Only participants receiving lopinavir/ritonavir capsules were planned to be followed past 9 months. | 36.4 (30.8) | NA (NA) — Only participants receiving lopinavir/ritonavir capsules were planned to be followed past 9 months.
  ALT - Baseline | 41.0 (40.3) | 39.6 (38.7) | 42.6 (42.6)
  ALT - 9 months | 39.8 (52.5) | 40.8 (44.8) | 39.0 (60.3)
  ALT - 18 months | NA (NA) — Only participants receiving lopinavir/ritonavir capsules were planned to be followed past 9 months. | 42.0 (44.8) | NA (NA) — Only participants receiving lopinavir/ritonavir capsules were planned to be followed past 9 months.

19. Primary Outcome: Laboratory Parameter Lipids
Description: A blood lipid panel consisting of total cholesterol, triglyceride, high-density lipoprotein (HDL), and low-density lipoprotein (LDL) levels was performed at baseline and scheduled study visits. Normal ranges are based on the standards for individual facilities in each country.
Time Frame: Baseline, 9 months, 18 months
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: millimoles per liter
Arm/Group | Total Study Population | Capsule Formulation | Tablet Formulation
Number analyzed (Participants) | 2288 | 1206 | 1016
millimoles per liter
  Total Cholesterol - Baseline | 4.37 (1.50) | 4.48 (1.68) | 4.28 (1.35)
  Total Cholesterol - 9 months | 4.96 (1.81) | 5.07 (2.36) | 4.89 (1.25)
  Total Cholesterol - 18 Months | NA (NA) — Only participants receiving lopinavir/ritonavir capsules were planned to be followed past 9 months. | 5.01 (1.29) | NA (NA) — Only participants receiving lopinavir/ritonavir capsules were planned to be followed past 9 months.
  HDL Cholesterol - Baseline | 1.39 (0.84) | 2.17 (1.45) | 1.19 (0.44)
  HDL Cholesterol - 9 months | 1.53 (0.98) | 2.08 (1.64) | 1.32 (0.53)
  HDL Cholesterol - 18 months | NA (NA) — Only participants receiving lopinavir/ritonavir capsules were planned to be followed past 9 months. | 2.04 (1.94) | NA (NA) — Only participants receiving lopinavir/ritonavir capsules were planned to be followed past 9 months.
  LDL Cholesterol - Baseline | 2.50 (1.07) | 2.87 (1.10) | 2.29 (1.02)
  LDL Cholesterol - 9 months | 2.73 (1.07) | 3.11 (1.18) | 2.51 (0.95)
  LDL Cholesterol - 18 months | NA (NA) — Only participants receiving lopinavir/ritonavir capsules were planned to be followed past 9 months. | 3.09 (1.14) | NA (NA) — Only participants receiving lopinavir/ritonavir capsules were planned to be followed past 9 months.
  Triglycerides - Baseline | 1.65 (1.06) | 1.66 (1.11) | 1.64 (1.04)
  Triglycerides - 9 months | 2.20 (1.46) | 2.21 (1.49) | 2.17 (1.44)
  Triglycerides - 18 months | NA (NA) — Only participants receiving lopinavir/ritonavir capsules were planned to be followed past 9 months. | 2.13 (1.35) | NA (NA) — Only participants receiving lopinavir/ritonavir capsules were planned to be followed past 9 months.

20. Secondary Outcome: Reasons for Discontinuation of Lopinavir/Ritonavir
Description: For participants who discontinued lopinavir/ritonavir treatment, the reasons for discontinuation are provided.
Time Frame: 9 months
Measure: Number; unit: Participants
Arm/Group | Total Study Population | Capsule Formulation | Tablet Formulation
Number analyzed (Participants) | 2288 | 1206 | 1016
Participants
  Number of participants discontinued | 269 | 122 | 143
  Lost to Follow-up | 167 | 61 | 104
  Adverse Event | 24 | 14 | 10
  Withdrawal by Subject | 7 | 6 | 1
  Treatment failure | 4 | 2 | 2
  Other - Tuberculosis/TB treatment | 4 | 4 | 0
  Other - Medication not available | 3 | 2 | 1
  Other - Poor general condition | 1 | 1 | 0
  Other - Increased triglycerides | 1 | 1 | 0
  Patient Noncompliance | 1 | 0 | 1
  Reason unknown | 57 | 31 | 24

21. Secondary Outcome: Reasons for Discontinuation of Lopinavir/Ritonavir
Description: For participants who discontinued lopinavir/ritonavir treatment, the reasons for discontinuation are provided.
Time Frame: 18 months
Population: Only participants receiving lopinavir/ritonavir capsules were planned to be followed past 9 months.
Measure: Number; unit: Participants
Arm/Group | Capsule Formulation
Number analyzed (Participants) | 1206
Participants
  Number of participants discontinued | 352
  Lost to Follow-up | 239
  Adverse Event | 20
  Withdrawal by Subject | 17
  Treatment failure | 7
  Other - Tuberculosis/TB treatment | 6
  Patient Noncompliance | 4
  Other - Medication not available | 3
  Other - Fatigue | 1
  Other - Increased triglycerides | 1
  Reason unknown | 54

22. Secondary Outcome: Compliance With Lopinavir/Ritonavir
Description: Participants reported whether they had missed doses of their antiretroviral treatment.
Time Frame: 9 months
Measure: Number; unit: Participants
Arm/Group | Total Study Population | Capsule Formulation | Tablet Formulation
Number analyzed (Participants) | 2288 | 1206 | 1016
Participants
  Reported never missing a dose | 1377 | 729 | 616
  Reported missing one or more doses | 853 | 459 | 361
  Information not reported | 58 | 18 | 39

23. Secondary Outcome: Compliance With Lopinavir/Ritonavir
Description: Participants reported whether they had missed any doses of their antiretroviral treatment.
Time Frame: 18 months
Population: Only participants receiving lopinavir/ritonavir capsules for followed for up to 18 months.
Measure: Number; unit: Participants
Arm/Group | Capsule Formulation
Number analyzed (Participants) | 1206
Participants
  Reported never missing a dose | 616
  Reported missing one or more doses | 578
  Information not reported | 12

24. Secondary Outcome: Adverse Events Observed on Treatment With Lopinavir/Ritonavir.
Description: Total number of adverse events with causal relationship (rated by Investigator as probably or possibly related) to lopinavir/ritonavir treatment.
  All serious adverse events and non serious adverse events (0.2% or greater frequency) are summarized in the "Reported Adverse Events" section of this record.
Time Frame: 18 months
Measure: Number; unit: Events
Arm/Group | Total Study Population | Capsule Formulation | Tablet Formulation
Number analyzed (Participants) | 2288 | 1206 | 1016
Events
  Total number of AEs with causal relationship | 260 | 175 | 78

ADVERSE EVENTS:
Time Frame: Study start through 9 months for all participants, and study start through 18 months for participants receiving lopinavir/ritonavir capsules.
Description: Adverse events (AEs) and Serious AEs occurring during the study were recorded. Serious AEs were reported from the time the physician obtained the patient's authorization to use and disclose information (or the patient's informed consent) until 30 days following intake of the last dose of the physician-prescribed lopinavir/ritonavir treatment.
Arm/Group | Total Study Population | Capsule Formulation | Tablet Formulation
Serious Adverse Events (participants affected / at risk) | 46/2288 | 22/1206 | 22/1016
Other Adverse Events (participants affected / at risk) | 109/2288 | 77/1206 | 34/1016
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Study Population (N=2288) | Capsule Formulation (N=1206) | Tablet Formulation (N=1016)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 1
Exophthalmos (Eye disorders) | 1 | 1 | 0
Iridocyclitis (Eye disorders) | 2 | 0 | 2
Mydriasis (Eye disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 3
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Asthenia (General disorders) | 1 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 1
Death (General disorders) | 7 | 2 | 5
Fatigue (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 3 | 3 | 0
Acquired immunodeficiency syndrome (Infections and infestations) | 2 | 2 | 0
Acute sinusitis (Infections and infestations) | 1 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 1 | 1
Cerebral toxoplasmosis (Infections and infestations) | 2 | 0 | 2
Encephalitis cytomegalovirus (Infections and infestations) | 1 | 0 | 1
Hepatitis C (Infections and infestations) | 1 | 1 | 0
Meningitis cryptococcal (Infections and infestations) | 1 | 1 | 0
Mycobacterium avium complex infection (Infections and infestations) | 2 | 0 | 2
Pharyngitis (Infections and infestations) | 1 | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 2 | 2 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0 | 1
Mycobacteria test (Investigations) | 1 | 1 | 0
Cachexiae (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 — Adverse event occurred in one of the 66 participants receiving both capsules and tablets, or oral solution.
Headache (Nervous system disorders) | 2 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 1 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 — One of the two adverse events occurred in one of the 66 participants receiving both capsules and tablets, or oral solution.
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Hospitalisation (Surgical and medical procedures) | 1 | 0 | 1
Thrombectomy (Surgical and medical procedures) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 0.2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total Study Population (N=2288) | Capsule Formulation (N=1206) | Tablet Formulation (N=1016)
Anaemia (Blood and lymphatic system disorders) | 4 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 8 | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 67 | 43 | 21 — One or more adverse events occurred in the 66 participants receiving both capsules and tablets, or oral solution.
Flatulence (Gastrointestinal disorders) | 3 | 3 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 4 | 1 | 3
Nausea (Gastrointestinal disorders) | 38 | 30 | 7 — One or more adverse events occurred in the 66 participants receiving both capsules and tablets, or oral solution.
Vomiting (Gastrointestinal disorders) | 24 | 17 | 6 — One or more adverse events occurred in the 66 participants receiving both capsules and tablets, or oral solution.
Asthenia (General disorders) | 10 | 6 | 4
Fatigue (General disorders) | 6 | 4 | 1 — One or more adverse events occurred in the 66 participants receiving both capsules and tablets, or oral solution.
Drug hypersensitivity (Immune system disorders) | 3 | 3 | 0
Weight decreased (Investigations) | 3 | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 | 5 | 1
Headache (Nervous system disorders) | 6 | 5 | 1
Depression (Psychiatric disorders) | 3 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.